CLINICAL TRIAL: NCT07243821
Title: Cohort Studies on Metabolic Syndrome and Prediabetes
Brief Title: Metabolic Syndrome and Prediabetes
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202509097RINB
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Metabolic Syndrome; Diabetes
Keywords: Obesity; Nutrition; Physical activity; Diabetes; Body composition; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to establish a cohort of individuals with metabolic syndrome and prediabetes to enable long-term follow-up of risk factors, disease progression, and the development of obesity-related complications. The study will also monitor changes in nutritional status and physical function over time, in order to identify key prognostic determinants influencing clinical outcomes.

Metabolic syndrome and prediabetes are chronic multisystem disorders, and poor long-term control is closely associated with the development of various complications. Moreover, malnutrition and functional decline are common comorbid conditions that further impair quality of life and impose a substantial burden on healthcare resources.

DETAILED DESCRIPTION:
Metabolic syndrome has been recognized as a significant contributor to the development of major chronic diseases, including cerebrovascular disorders, cardiovascular disease, diabetes mellitus, and hypertension. Compared with the general population, individuals with metabolic syndrome exhibit an approximately sixfold increased risk of diabetes, fourfold risk of hypertension, threefold risk of dyslipidemia, and twofold risk of stroke and coronary heart disease.

The condition is strongly influenced by dietary and lifestyle factors. Its core pathophysiological features are insulin resistance and central obesity, and there is a high degree of comorbidity between metabolic syndrome and prediabetes.

The establishment of a comprehensive cohort and database for individuals with metabolic syndrome and prediabetes will facilitate the systematic collection of metabolic profiles and disease-related biomarkers. This will enable longitudinal analyses of systemic and organ-specific complications, their incidence, and predictive determinants, thereby strengthening disease risk stratification and early identification.

This study aims to collect routine clinical, physiological, and nutritional data at regular intervals to examine associations among lifestyle behaviors, metabolic factors, physiological indicators, and the development of complications. Furthermore, it seeks to evaluate nutritional and functional status, identify potential prognostic biomarkers, and provide a foundation for individualized therapeutic approaches and integrated healthcare models.

ELIGIBILITY:
Inclusion Criteria

1. Adults aged 18 years or older.
2. Individuals clinically diagnosed by a physician as having metabolic syndrome (meeting at least three of the following five criteria) or prediabetes:

   (A) Waist circumference: ≥ 90 cm in men or ≥ 80 cm in women, or body mass index (BMI) ≥ 27 kg/m².

   (B) Fasting plasma glucose (AC): ≥ 100 mg/dL. (C) Blood pressure: Systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmHg.

   (D) Triglycerides (TG): ≥ 150 mg/dL. (E) High-density lipoprotein cholesterol (HDL-C): < 40 mg/dL in men or < 50 mg/dL in women.
3. Individuals meeting the definition of prediabetes, defined as glycated hemoglobin (HbA1c) between 5.7% and 6.4%.
4. Participants who are willing to participate in the study and have signed written informed consent.
5. Participants who are able to complete basic physical examinations and assessment procedures.

Exclusion Criteria

1. Individuals unable to comprehend the study information or procedures.
2. Individuals unable to comply with the required assessments or study protocols.
3. Any other condition that, in the clinical judgment of the principal investigator, deems the individual unsuitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: articipants eligible for inclusion are adults aged 18 years or older who have been clinically diagnosed with either metabolic syndrome or prediabetes. Metabolic syndrome is defined by the presence of at least three of the following five criteria: (A) waist circumference ≥ 90 cm in men or ≥ 80 cm in women, or a body mass index (BMI) ≥ 27 kg/m²; (B) fasting plasma glucose ≥ 100 mg/dL; (C) systolic blood pressure ≥ 130 mmHg or diastolic blood pressure ≥ 85 mmHg; (D) triglycerides ≥ 150 mg/dL; and (E) high-density lipoprotein cholesterol (HDL-C) < 40 mg/dL in men or < 50 mg/dL in women.
  Participants meeting the definition of prediabetes, defined as glycated hemoglobin (HbA1c) levels between 5.7% and 6.4%, will also be eligible. All participants must be willing to join the study, provide written informed consent, and be able to complete basic physical examinations and assessment procedures.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Medical record system and on-site inspection data collection | Everytime after physician's appointment(Usually 3 months).

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Wen Lu, Present Professor, Study Chair — Department of Family Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided